CLINICAL TRIAL: NCT07362030
Title: A Open-Label, Phase I Drug-drug Interaction Clinical Study to Investigate the Pharmacokinetics of RAY1225 With Warfarin, Atorvastatin, Metformin and Digoxin in Healthy Participants
Brief Title: Drug-durg Interaction of RAY1225 With Warfarin, Atorvastatin, Metformin and Digoxin
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RAY1225-24-11
Record Dates: First submitted 2026-01-14; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Atorvastatin; Metformin; Warfarin; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental 1 (Experimental): Period 1: All participants took one tablet of atorvastatin calcium (20mg) and one tablet of metformin hydrochloride (500mg) in the morning of Day 1, after fasting. On the morning of Day 8, they took two tablets of warfarin sodium (5mg) and one tablet of digoxin (0.25mg) in the same fasting condition.
  Period 2: All participants were injected with RAY1225 once every two weeks (a total of 7 times, with each dose ranging from 1mg to 3mg to 6mg to 6mg to 6mg to 6mg to 6mg). On D86 (24±1 hours after the 6th administration of RAY1225), they took 1 tablet of atorvastatin calcium (20mg) and 1 tablet of metformin hydrochloride (500mg) orally in an empty stomach condition with approximately 240ml of warm water. On D100 (24±1 hours after the 7th administration of RAY1225), they took 2 tablets of warfarin sodium (5mg) and 1 tablet of digoxin (0.25mg) orally in an empty stomach condition with approximately 240ml of warm water in the morning.
  Interventions: Drug: RAY1225; Drug: atorvastatin calcium tablet; Drug: Metformin Tablets; Drug: Warfarin Sodium Tablets; Drug: Digoxin Tablets

INTERVENTIONS:
Drug: RAY1225 — subcutaneous injection
Drug: atorvastatin calcium tablet — Oral
Drug: Metformin Tablets — Oral
Drug: Warfarin Sodium Tablets — Oral
Drug: Digoxin Tablets — Oral

SUMMARY:
The drug-drug interaction study had been designed to investigate the effect of RAY1225 on the pharmacokinetics of digoxin, Rosuvastatin and

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) ≥20 to ≤35 kg/m2 and total body weight >50 kg(male) or >45kg(female) at Screening (calculated as a function of measured height and weight according to the formula, BMI = kg / m2 where m2 is height in meters squared);
2. Ability to understand and willingness to sign a written informed consent form;
3. Normal physical examination, vital signs, 12-lead ECG, and clinical laboratory values, or any abnormality that is non-clinically significant.

Exclusion Criteria:

1. Participants with a history of hypersensitivity to study drug or any component of study medication;
2. Participants had taken prescription, over-the-counter, herbal, or vitamin products within 4 weeks prior to screening；
3. Smoking more than 5 cigarettes per day within 12 weeks prior to screening，or who cannot stop using any tobacco products during the study period;
4. Participants who donated blood/bleeding profusely (> 400 mL) 12 weeks prior to randomization;
5. Those with clinically significant Electrocardiogram(ECG) abnormalities, or QTcF > 450ms;
6. Participants who test positive at Screening and/or admission (Day -1) for alcohol abuse.
7. Females who are pregnant, lactating, or likely to become pregnant during the study.
8. History of dysphagia or any gastrointestinal disorder that affect absorption

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2025-04-14 (Actual); Primary Completion 2025-12-27 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic - Cmax | Day 1~Day 5 and Day 86~Day 107
  Maximum observed plasma concentration
Pharmacokinetic -Area under the curve（AUC） | Day 1~Day 5 and Day 86~Day 107
  Area under the curve

SECONDARY OUTCOMES:
Number of participants with adverse events | DAY 1~Day 107
  The safety and tolerability of RAY1225 alone and in combination with IWarfarin, atorvastatin, metformin and digoxin will be examined.

CONTACTS AND LOCATIONS:
Locations (1):
- Dongguan People's Hospital, Dongguan, China